CLINICAL TRIAL: NCT06998212
Title: The Effect of Smartphone-Based Recording Offer on Patient Satisfaction in Orthopedic Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Blake Han (Other)
Collaborators: Riverside University Health System Medical Center (Other)
Responsible Party: Sponsor-Investigator, Blake Han, Research Coordinator, Riverside University Health System Medical Center
Organization: Riverside University Health System Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2327150-1
Record Dates: First submitted 2025-05-19; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Patient Satisfaction
Keywords: Satisfaction; Smartphone; Recording; Record; Preop; Preoperative; Orthopedic
MeSH Terms: conditions — Patient Satisfaction; Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Offer to record the encounter on patient smartphone (Experimental)
  Interventions: Behavioral: Offer to record encounter
- No offer to record the encounter on patient smartphone (No Intervention)

INTERVENTIONS:
Behavioral: Offer to record encounter — Patient will be given the option to record their clinical encounter on their personal smartphone
  Arms: Offer to record the encounter on patient smartphone

SUMMARY:
The purpose of this study is to determine patient satisfaction with orthopedic preoperative encounter based on offer to record the encounter on patient personal smartphone.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting to RUHS for preoperative orthopedic evaluation

Exclusion Criteria:

* Patients without smartphones

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 972 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction with preoperative orthopedic encounter | From enrollment to survey completion
  Measured via survey response

SECONDARY OUTCOMES:
Patient survey responses including if patient recorded visit, reason for recording visit, preference for recording visit | From enrollment to survey completion
  Survey Responses
If satisfaction varies by demographic factors (age, race, ethnicity, sex) or by type of procedure that the preop is for | Through study completion, average 1 year
  Information will be collected from chart review

CONTACTS AND LOCATIONS:
Locations (1):
- Riverside University Health System, Moreno Valley, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Demographics, reason for encounter, survey responses
Supporting Information: Study Protocol, ICF
Access Criteria: No plans to share data at this time.

REFERENCES:
- [Background] Norgaard B, Kofoed PE, Ohm Kyvik K, Ammentorp J. Communication skills training for health care professionals improves the adult orthopaedic patient's experience of quality of care. Scand J Caring Sci. 2012 Dec;26(4):698-704. doi: 10.1111/j.1471-6712.2012.00982.x. Epub 2012 Mar 16. PMID 22420418
- [Background] Meakin R, Weinman J. The 'Medical Interview Satisfaction Scale' (MISS-21) adapted for British general practice. Fam Pract. 2002 Jun;19(3):257-63. doi: 10.1093/fampra/19.3.257. PMID 11978716
- [Background] Koh TH, Butow PN, Coory M, Budge D, Collie LA, Whitehall J, Tattersall MH. Provision of taped conversations with neonatologists to mothers of babies in intensive care: randomised controlled trial. BMJ. 2007 Jan 6;334(7583):28. doi: 10.1136/bmj.39017.675648.BE. Epub 2006 Dec 1. PMID 17142256
- [Background] Wolderslund M, Kofoed PE, Holst R, Axboe M, Ammentorp J. Digital audio recordings improve the outcomes of patient consultations: A randomised cluster trial. Patient Educ Couns. 2017 Feb;100(2):242-249. doi: 10.1016/j.pec.2016.08.029. Epub 2016 Aug 29. PMID 27593087
- [Background] Elwyn G, Barr PJ, Grande SW. Patients recording clinical encounters: a path to empowerment? Assessment by mixed methods. BMJ Open. 2015 Aug 11;5(8):e008566. doi: 10.1136/bmjopen-2015-008566. PMID 26264274